CLINICAL TRIAL: NCT01271946
Title: A Patient Registry Evaluating Closure Following Access With the ArstasisOne Access System
Acronym: RECITAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arstasis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-03133
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Results first posted 2013-01-17 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Diagnostic Catheterization Access Through a 5F or 6F Femoral Artery Introducer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic Procedure (Other)
  Interventions: Device: Diagnostic catheterization procedure

INTERVENTIONS:
Device: Diagnostic catheterization procedure — Intervention includes diagnostic catheterization procedure involving access through a 5F or 6F introducer in the femoral artery.

SUMMARY:
The goal of this study is to observe the clinical safety and effectiveness of the ArstasisOne Access System in patients undergoing diagnostic angiographic procedures through the femoral artery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 85 years of age.
* Patient is clinically indicated for a diagnostic catheterization procedure involving access through a 5F or 6F introducer in the femoral artery.
* Patient is able to ambulate without assistance prior to the procedure and can be expected to ambulate (20 feet) post-procedure.

Exclusion Criteria:

* Patient is unable to routinely walk at least 20 feet without assistance (e.g., requires a walker or wheelchair to mobilize or has known paralysis).
* Patient has an active systemic or cutaneous infection or inflammation (e.g., septicemia at the time of the procedure).
* Patient has systemic hypertension unresponsive to treatment (>180mmHg systolic and >110mmHg diastolic).
* Patient has received thrombolytic therapy within the 72 hours prior to catheterization.
* Patient has a previously diagnosed significant bleeding coagulopathy, is on warfarin and has an INR ≥ 1.5 or has a platelet disorder, including known thrombocytopenia (platelet count <100,000), thrombasthenia, Von Willebrand's disease, Factor V deficiency, or anemia (Hemoglobin< 10 g/dL, or Hct<30%).
* Patient has a compromised femoral artery access site.
* Patient procedure requires an introducer sheath size of> 6F.
* Patient has had prior vascular surgery or vascular grafts at the femoral artery access site.
* Patient presents with hemodynamic instability or is in need of emergent surgery.
* Patient has received femoral artery closure on the target access vessel with a collagen/PEG closure device within 90 days of the current procedure.
* Patient has a pre-existing severe non-cardiac systemic disease or illness that results in an expected life expectancy of< 30 dys or for other reasons has a life expectancy of less than 1 yaer.
* Patient is currently participating in an investigational drug or another device study that clinically interferes with the current study endpoints.
* Pregnant or lactating patients.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zoltan Turi, MD, Principal Investigator — The Cooper Health System; John Held, MD, Principal Investigator — Mercy Hospital Fairfield; Frank Kresock, MD, Principal Investigator — The Cardiovascular Center; Tom Hinohara, MD, Principal Investigator — Sequoia Hospital; Dale Wortham, MD, Principal Investigator — Volunteer Research Group, LLC; Greg Sampognaro, MD, Principal Investigator — P&S; Ray Smith, MD, Principal Investigator — Ark-La-Tex Cardiology/Willis-Knighton Hospital; Kalyan Veerina, MD, Principal Investigator — Cardiovascular Institute of the South-Opelousas
Locations (8):
- United States (8):
  - The Cardiovascular Center, Parker, Arizona
  - Sequoia Hospital, Redwood City, California
  - P&S Surgical Hospital, Monroe, Louisiana
  - Cardiovascular Institute of the South-Opelousas, Opelousas, Louisiana
  - Willis-Knighton Hospital, Shreveport, Louisiana
  - The Cooper Health System, Camden, New Jersey
  - Mercy Hospital Fairfield, Fairfield, Ohio
  - Volunteer Research Group, LLC, Knoxville, Tennessee

REFERENCES:
- [Derived] Turi ZG, Wortham DC, Sampognaro GC, Kresock FD, Held JS, Smith RD, Veerina KK, Hinohara T, Kaki A. Use of a novel access technology for femoral artery catheterization: results of the RECITAL trial. J Invasive Cardiol. 2013 Jan;25(1):13-8. PMID 23293169

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment commenced November 3, 2010 and concluded June 3, 2011. Patients who underwent routine diagnostic catheterization through 5 or 6F sheaths were enrolled in the study at 8 investigational sites in the US.
Pre-assignment Details: Patients were required to be able to ambulate without assistance prior to the procedure and can be expected to ambulate (20 feet) post-procedure.
Groups:
- Intent to Treat (ITT): The ITT cohort consists of those subjects where an attempt was made to place the Arstasis device into subject's vasculature regardless of whether or not this attempt was successful.
- Sheath Greater Than 6 French (F): Subjects in whom the procedural sheath was upsized to greater than 6F.
Period: Overall Study
Arm/Group | Intent to Treat (ITT) | Sheath Greater Than 6 French (F)
Started | 346 | 5
Completed | 346 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intent to Treat | Sheath Greater Than 6F | Total
Number analyzed (Participants) | 346 | 5 | 351
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 161 | 4 | 165
  >=65 years | 185 | 1 | 186
Age Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.8) | 63.2 (11.7) | 64.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 2 | 153
  Male | 195 | 3 | 198
Region of Enrollment [Number; unit: participants]
  United States | 346 | 5 | 351

OUTCOME MEASURES:

1. Primary Outcome: Observation of Any Site Related Complications Recorded as Either Major or Minor Adverse Events.
Time Frame: Procedure through 30 days follow-up.
Reporting Status: Not Posted

2. Primary Outcome: Major Adverse Events Reported as Percentage of Participants With Adverse Events.
Description: Observation of any major access site-related complication (percentage of participants).
Time Frame: Procedure through 30 day follow-up.
Measure: Number; unit: Percentage of participants
Groups:
- Intent to Treat: Major access site-related complications observed in the intent-to-treat population.
- Sheath Greater Than 6F: Major access site-related complications observed in subjects treated with sheath size greater than 6F.
Arm/Group | Intent to Treat | Sheath Greater Than 6F
Number analyzed (Participants) | 346 | 5
Percentage of participants | 0 | 0

3. Primary Outcome: Device Success
Description: Achievement of femoral artery access using the Arstasis Access System followed by placement of the procedural sheath in the femoral artery.
Time Frame: Procedure
Population: Intent to treat.
Measure: Number; unit: Percentage of participants
Arm/Group | Intent to Treat | Sheath Greater Than 6F
Number analyzed (Participants) | 346 | 5
Percentage of participants | 97 | 100

4. Primary Outcome: Minor Adverse Events
Description: Observation of any minor access site-related complications.
Time Frame: Procedure through 30 day follow-up.
Measure: Number; unit: Percentage of participants
Groups:
- Group 1: Minor access site-related complications observed in the intent-to-treat population.
- Sheath Greater Than 6F: Minor access site-related complications observed in subjects who were upsized to sheath size greater than 6F.
Arm/Group | Group 1 | Sheath Greater Than 6F
Number analyzed (Participants) | 346 | 5
Percentage of participants | 4.0 | 0

5. Primary Outcome: Time to Hemostasis
Description: The difference between the time the procedural sheath was removed from the femoral artery and the time when hemostasis was observed.
Time Frame: Hemostasis was evaluated immediately following procedural sheath removal until hemostasis was achieved.
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Intent to Treat; Sheath Greater Than 6F: Time to Hemostasis was evaluated in subjects in whom successful acess with the Arstasis device was achieved and data was available.
Arm/Group | Intent to Treat | Sheath Greater Than 6F
Number analyzed (Participants) | 334 | 4
Minutes | 4.8 (3.7) [4.4 to 5.2] | 6.0 (4.2)

6. Primary Outcome: Time to Discharge Eligibility
Description: The time from sheath removal to the time when the subject was medically able to be discharged based solely on the assessment of the access site.
Time Frame: Discharge Eligibility was evaluated following sheath removal and ambulation and physical examination of the access site demonstrating stable access site.
Population: Per Protocol.
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Group 1: Time to Discharge Eligibility was evaluated in subjects in whom successful acess with the Arstasis device was achieved and data was available.
Arm/Group | Group 1 | Sheath Greater Than 6F
Number analyzed (Participants) | 333 | 4
Hours | 6.0 (7.6) | 10.7 (9.9)

7. Primary Outcome: Time to Actual Discharge
Description: The time from sheath removal to actual hospital discharge.
Time Frame: Actual discharge was evaluated following procedural sheath removal until actual discharge, an average time of 9.3 hours.
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Intent to Treat: Time to Actual Discharge was evaluated in subjects in whom successful acess with the Arstasis device was achieved and data was available.
Arm/Group | Intent to Treat | Sheath Greater Than 6F
Number analyzed (Participants) | 335 | 4
Hours | 9.3 (22.1) | 12.8 (11.8)

8. Primary Outcome: Time to Ambulation
Description: Time to ambulation was recorded as the difference between the time the procedural sheath is removed from the femoral artery and the time when the subject stands and walks at least 20 feet without re-bleeding.
Time Frame: Ambulation was evaluated at any time after 1, 2 and 4 hours post sheath removal, until the subject was successfully ambulated.
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Intent to Treat; Sheath Greater Than 6F: Time to Ambulation was evaluated in subjects in whom successful acess with the Arstasis device was achieved and data was available.
Arm/Group | Intent to Treat | Sheath Greater Than 6F
Number analyzed (Participants) | 332 | 4
Hours | 2.0 (2.1) | 1.8 (0.5)

9. Primary Outcome: Percentage of Participants With Bed Elevation Within 15 Minutes.
Description: Successful bed elevation was defined as the ability to sit up at a 45 degree angle within 15 minutes (1-30 minutes window) following sheath removal and successful hemostasis, without re-bleeding. This outcome was evaluated in subjects in whom successful access with the Arstasis device was achieved. The outcome measurement is reported as percentage of subjects.
Time Frame: Post procedure
Population: Per protocol.
Measure: Number; unit: Percentage of participants
Groups:
- Intent to Treat; Sheath Greater Than 6F: Time to Bed Elevation was evaluated in subjects in whom successful access with the Arstasis device was achieved and data was available.
Arm/Group | Intent to Treat | Sheath Greater Than 6F
Number analyzed (Participants) | 245 | 1
Percentage of participants | 99.6 | 20

10. Secondary Outcome: Time to Hemostasis
Description: Time to hemostasis for the diagnostic cohort, compared to published literature rates of 17 minutes for time to hemostasis for standard manual compression.
Time Frame: Hemostasis was evaluated immediately following procedural sheath removal.
Population: Per protocol-Diagnostic Cohort.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Per Protocol: Time to Hemostasis was evaluated in subjects in whom successful acess with the Arstasis device was achieved and data was available.
Arm/Group | Per Protocol
Number analyzed (Participants) | 241
Minutes | 4.0 (2.5)

11. Secondary Outcome: Time to Ambulation
Description: Time to ambulation for the diagnostic cohort, compared to published literature rates of 4.75 hours for time to ambulation for standard manual compression.
Time Frame: as for outcome 8
Population: Per Protocol-Diagnostic Cohort.
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Per Protocol: Time to Ambulation was evaluated in subjects in whom successful access with the Arstasis device was achieved and data was available.
Arm/Group | Per Protocol
Number analyzed (Participants) | 240
Hours | 1.5 (1.2)

ADVERSE EVENTS:
Time Frame: Procedure through 30 day post procedure.
Arm/Group | Intent to Treat | Sheath Greater Than 6F
Serious Adverse Events (participants affected / at risk) | 0/346 | 0/5
Other Adverse Events (participants affected / at risk) | 0/346 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission for publication or presentation, the Institution will provide the Sponsor with at least sixty (60) days for review of a manuscript. If requested in writing,The Institution and Principal Investigator will withhold such publication for up to an additional sixty (60) days to allow for filing of a patent application.